CLINICAL TRIAL: NCT01799070
Title: Velocity Systolic Blood Pressure Index in Accurately Predicting Cerebral Hyperperfusion Syndrome After Carotid Endarterectomy
Brief Title: Accuracy of TCD Monitoring in Predicting Cerebral Hyperperfusion Syndrome After Carotid Endarterectomy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Liu Bao, M.D., Peking Union Medical College Hospital
Other Study IDs: PUMCH-20130113; B2009B080 (Other Grant/Funding Number: Central Committee of China health care Administration)
Record Dates: First submitted 2013-02-24; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Carotid Stenosis; Cerebral Hyperperfusion Syndrome; Blood Pressure
Keywords: Prediction; Transcranial Doppler
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CHS

SUMMARY:
Background: Cerebral hyperperfusion syndrome (CHS) is a life threatening complication of carotid endarterectomy (CEA) and the changes of middle cerebral artery velocity are used to predict the occurrence of CHS but the accuracy is limited. In addition, changes of BP post-operatively comparing with baseline BP should be a predictive factor of CHS.

Objective: The investigators aimed to create a predictive index, velocity systolic blood pressure index (VSI), for improving the predictive power of Transcranial Doppler monitoring regarding CHS.

Methods: The study design is a diagnostic test, which is an observational analytic clinical study. From March 2013 to September 2014, 200 patients will be recruited. Patients will be classified according to the CHS occurrence. VSI combined the changes of middle cerebral artery velocity and blood pressure crossing CEA and the intra- and post-operative increase ratios of middle cerebral artery velocity were calculated. Their prediction power of CHS will be compared. Sensitivity, specificity, positive predictive value, negative predictive value of them will be calculated. Receiver operating characteristic analysis will be performed.

Expected Outcomes: Comparing with the commonly used intra-operative and post-operative TCD monitoring, VSI may be more useful to select CHS in patients who underwent CEA. As far as the investigators know, analysis or studies combining the BP and velocity changes in the prediction of CHS have never been performed.

DETAILED DESCRIPTION:
This study is designed as a standard diagnostic test. It is designed to verify the predictive power of VSI with CHS, and which is an observational analytic clinical study. The investigative parameters of patients will be collected prospectively by the designed case report form. According to the incidence of CHS, the estimated enrollment amount is set as 200. Patients will be recruited by the inclusion and exclusion criteria below. All the patients included will accept the standard CEA surgery treatment in the department of vascular surgery of PUMCH. MCAV and systolic BP data will be recorded cross CEA. Post-operatively the CHS patients will be identified according to the golden standard. The golden standard is the clinical diagnose of CHS (the detailed diagnostic criteria will be stated in the methodology part). The TCD operator is blind to the patients. The predictive power of VSI will be identified by the sensitivity, specificity, positive predictive value, negative predictive value and ROC plot comparing with the golden standard. The study start date is March 2013, the estimated study completion date is December 2014 and the primary completion date is September 2014 (final data collection date for primary outcome measure).

ELIGIBILITY:
Inclusion Criteria:

1. Age from 30 to 85 years;
2. Had a middle-grade symptomatic carotid stenosis (more than 50%) or a high-grade asymptomatic carotid stenosis (more than 70%);
3. Underwent CEA 30 days after the last ischemic cerebrovascular event in the case of symptomatic carotid stenosis;
4. Signed the ethical information consent form
5. Underwent TCD study intraoperative and immediately after CEA;
6. The degree of carotid stenosis will be assessed by CT angiography or cerebral digital subtraction angiography (DSA). (The method document came from the North American Symptomatic Carotid Endarterectomy Trial study.)

Exclusion Criteria:

1. Emergency CEA within 30 days of stroke onset in the case of symptomatic carotid stenosis;
2. No temporal windows to measure the MCAV.
3. Restenosis after CEA or CAS
4. Stenosis caused by non-atherosclerotic diseases
5. Combined severe systematic diseases that markedly decrease the life cycle
6. Allergy to medicines of the study such as Aspirin or Statin
7. Refuse to sign the ethical information consent form

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who with carotid stenosis will accept CEA in PUMCH from March 2013 to September 2014.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
cerebral hyperperfusion syndrome | within 7 days after surgery
  CHS will be diagnosed if (1) the patient developed symptoms that ipsilateral moderate or severe headache, confusion, seizures, intracranial hemorrhage or focal neurological deficits after a symptom-free interval. (2) symptoms not secondary to cerebral ischemia which will be excluded by CT or MRI. (3) MCAV increasing >100% from baseline which identified by TCD. (4) within 7 days after surgery. (5) An independent neurologist made the diagnosis of CHS.

CONTACTS AND LOCATIONS:
Locations (1):
- vascular surgery department of PUMCH, Beijing, Beijing Municipality, China